CLINICAL TRIAL: NCT01684618
Title: Oxygenation of the Neonatal Brain - a Study Using the INVOS Oximeter
Brief Title: Neonatal Cerebral Oxygenation and Changes in CPAP Flow Pressure - Evaluation With INVOS Oximeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: The Ludvig & Sara Elsass Foundation (Unknown)
Responsible Party: Principal Investigator, Line Carøe Sørensen, MD, PH.D., Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CPAP - HH 527
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Cerebral Oxygenation
Keywords: Preterm; Neonate; Newborn; Cerebral oxygenation; CPAP
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cerebral NIRS oximetry + CPAP (Experimental): Cerebral NIRS oximetry, using the INVOS Cerebral/Somatic Oximeter, and changes in regional cerebral oxygen saturation, rSO2, during induced changes in CPAP flow pressure
  Interventions: Procedure: Cerebral NIRS Oximetry + CPAP

INTERVENTIONS:
Procedure: Cerebral NIRS Oximetry + CPAP — CPAP flow pressure is increased for 5 minutes then 15 minutes with CPAP pressure at baseline. Repeated once
  Other Names: INVOS 5100C Oximeter

SUMMARY:
* Due to the increased risk of brain damage, continuous monitoring of the cerebral oxygenation is interesting. We will evaluate the capability of the INVOS Oximeter to detect induced changes in the cerebral regional saturation.
* The purpose of the study is to investigate our hypothesis that a particular CPAP flow pressure optimizes the regional cerebral oxygenation.

DETAILED DESCRIPTION:
Preterm infants are at increased risk of brain damage compared with term infants, and cerebral hypoxia is considered to have an important role. The preterm infants are at increased risk of respiratory distress, episodes with low oxygenation, mechanical ventilation, risk of hypocapnia and labile or low blood pressure. These conditions can affect the microcirculation and hence the oxygenation of the brain. Hyperoxia is also a point of interest, since high levels of oxygen can cause vasoconstriction. Preterm infants is often treated with CPAP (Continuous positive airway pressure), but the effect of different flow pressures on the regional cerebral oxygenation is not known.

The investigators will examine the normal physiological response of the brain in a group of preterm infants with a gestational age (GA) of 32-37 weeks and a group of term infants to the commonly used treatment in neonatology, CPAP (Continuous positive airway pressure).

The investigators will do dynamic research with continuously monitoring of the cerebral oxygenation using the INVOS® Cerebral/Somatic Oximeter (Near InfraRed Spectroscopy (NIRS)). INVOS® is the first NIRS-based oximeter CE-approved for hospital use in Denmark.

There will be no follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: - Newborns with a gestational age of 32-40 weeks - Clinically stable - +/- CPAP with a oxygen limit below 30% - Parental consent

Exclusion Criteria:

* Severe birth asphyxia - Prohibition of oxygen exposure

Ages: 1 Hour to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in regional cerebral oxygen saturation, rSO2, during induced changes in CPAP flow pressure | Measurements will take between 30 minutes and 3 hours depending of situation. Within the first 4 weeks of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, Copenhagen University Hospital; Hvidovre, Hvidovre, Denmark